CLINICAL TRIAL: NCT05070988
Title: Oral Health Related Quality of Life of Patients With Rare Diseases Followed at Necker Hospital: a Qualitative Approach
Brief Title: Oral Health Related Quality of Life of Patients With Rare Diseases: a Qualitative Approach
Acronym: RaroDentAXE3
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210890; 2021-A00429-32 (Other: ID RCB number)
Record Dates: First submitted 2021-09-27; First posted 2021-10-07 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Rare Diseases
Keywords: Rare diseases; Oral health-related quality of life; Qualitative method
MeSH Terms: conditions — Rare Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Rare diseases: Children and adult patients with rare diseases and followed at the Necker Enfant Malades Hospital, Paris
  Interventions: Other: Semi-structured interview

INTERVENTIONS:
Other: Semi-structured interview — Semi-structured interview with the investigating doctor of the study lasting 30 minutes to an hour

SUMMARY:
The main objective of the study is to assess the oral health-related quality of life of patients with rare diseases and followed in the rare disease centers of expertise at Necker Hospital in Paris by semi-structured interviews.

DETAILED DESCRIPTION:
To date, few studies have used the qualitative method to analyze the oral health-related quality of life and the oral health care pathways of patients with rare diseases, all health sectors combined. The quantitative studies carried out using standardized questionnaires offer only a partial view of how patients feel, both children and adults.

The main objective of the study is to assess the oral health-related quality of life of patients with rare diseases and followed in the rare disease centers of expertise at Necker Hospital in Paris by means of a semi-structured interview.

ELIGIBILITY:
Inclusion Criteria:

* Minor and adult patients with rare diseases aged of at least 6 years old and followed at the Necker Enfant Malades Hospital, Paris
* Patients with the 3 most frequent rare diseases of each rare disease Necker reference center participating in the study (10 centers : Chronic And Malformative Disorders Of The Esophagus / Inflammatory diseases of the bile ducts and autoimmune hepatitis / Constitutional Bone Diseases / Inherited Metabolic Diseases / Biliary Atresia And Genetic Cholestases / Vascular Diseases Of The Liver / Developmental Anomalies and Malformative Syndromes of Ile-De-France / Rare Causes Intellectual Disabilities / Complex congenital heart defects / Childhood cerebrovascular pathologies)
* Patients who consulted between 1.1.2017 and 1.1.2020 the relevant rare disease reference center at Necker hospital
* Patients seen at least once in the medical genetics department of Necker Hospital
* Information and non-opposition of adult patients / holders of parental authority of minor patients and minor patients to participate in the study

Exclusion Criteria:

Patients who do not speak French

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is that of the centers of expertise for rare diseases at the Necker Hospital in Paris, France.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2021-11-29 (Actual)

PRIMARY OUTCOMES:
Oral health-related quality of life assessment | Day 0
  Qualitative method from a semi-structured interview.

SECONDARY OUTCOMES:
Description of oral health care pathways | Day 0
  Description from the semi-structured interviews.
Inequalities in access to oral health care | Day 0
  Description of inequalities in access to oral health care. Description from the semi-structured interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Friedlander, DDS, PHD, associate professor, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Friedlander L, Berdal A, Cormier-Daire V, Lyonnet S, Garcelon N. Determinants of dental care use in patients with rare diseases: a qualitative exploration. BMC Oral Health. 2023 Jun 22;23(1):413. doi: 10.1186/s12903-023-03048-1. PMID 37349716